CLINICAL TRIAL: NCT02593253
Title: The Effect of a Novel Electronic Physician Audit and Feedback Bundle on Inpatient Performance Metrics
Brief Title: The Effect of a Novel Audit and Feedback Bundle on Inpatient Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-17709
Record Dates: First submitted 2015-10-23; First posted 2015-11-02 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Quality Improvement
Keywords: Quality Improvement; Quality Indicators, Health Care; Hospital Medicine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Audit and Feedback Bundle (Experimental): Access to the electronic dashboard and weekly feedback rounds
  Interventions: Other: Audit and Feedback Bundle
- Bi-weekly audit and feedback emails (Active Comparator): Access to biweekly feedback emails with performance on selected quality measures (current practice).
  Interventions: Other: Bi-weekly audit and feedback emails

INTERVENTIONS:
Other: Audit and Feedback Bundle — The intervention arm teams will receive the new audit and feedback bundle, which includes access to the electronic dashboard and weekly feedback rounds in which they review their performance on several inpatient quality metrics via the dashboard.
  Arms: Intervention Audit and Feedback Bundle
Other: Bi-weekly audit and feedback emails — The control arm will undergo audit and feedback per the current system, which is biweekly feedback emails with performance on selected quality measures.
  Arms: Bi-weekly audit and feedback emails

SUMMARY:
This single-blinded, cluster randomized control trial will assess the effectiveness of an audit and feedback bundle on internal medicine physician performance on selected quality metrics. The feedback bundle includes an electronic dashboard and weekly feedback rounds in which physicians will review their performance. The control arm will undergo audit and feedback per the current system, which is biweekly feedback emails with performance.

DETAILED DESCRIPTION:
This is a single-blinded, cluster randomized control trial of 48 internal medicine teams (24 teams will be randomized to the intervention arm and and 24 teams randomized to control arm) on inpatient medicine wards. Each team consists of at least 4 members (attending physician, senior resident, two interns). The intervention arm teams will receive the new audit and feedback bundle, which includes access to the electronic dashboard and weekly feedback rounds in which they review their performance on several inpatient quality metrics via the electronic dashboard. The control arm will undergo audit and feedback per the current system, which is biweekly feedback emails with performance on selected quality measures. This primary aim of the trial will be to compare the effectiveness of performance feedback on inpatient quality metrics specifically high quality after visit summary, medical reconciliation and discharge summary timeliness. Other group comparisons will include other inpatient quality metrics and satisfaction with feedback.

ELIGIBILITY:
Inclusion Criteria:

* All physicians that rotate through internal medicine wards during the study period (teaching attending physicians and internal medicine residents and interns)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a high quality after visit summary | 6 months
  The number of hospital medicine team patients with after visit summaries of high quality divided by the total number hospital medicine team patients with an after visit summary.
Proportion of patients with discharge summary timeliness | 6 months
  The number of discharge summaries completed within 24 hours of discharge for hospital medicine team patients/total number of discharges from hospital medicine with a discharge summary completed
Proportion of patients Complete Medication Reconciliation by Discharge | 6 months
  The total number of patients with an action taken on all home medications divided by the total number of patients on the hospital medicine teaching service.
Proportion of patients achieving a high quality 'perfect' discharge | 6 months
  Proportion of patients who have a high quality after visit summary and a discharge summary completed within 24 of discharge and all medications reconciled by discharge.

SECONDARY OUTCOMES:
Proportion of attending and resident physicians who 'strongly agree' that they are satisfied with the audit and feedback of performance data that they receive. | 6 months
  Proportion of attending and resident physicians who 'strongly agree' that they are satisfied with the audit and feedback of performance data that they receive. This specific satisfaction item has been developed by the study team.
Total Phlebotomy Sticks | 6 months
  The total number of unique accession numbers for each unique hospitalization of a patient
Percent of Patients on Telemetry Until Discharge | 6 months
  The number of patients on without a discontinue order for telemetry within two hours of their discharge date time divided by the total number of patients on telemetry for hospital medicine teams
Proportion of patients discharged by noon | 6 months
  The number of patients discharged by hospital medicine team attendings by noon (6am-11:59am)/total number of discharges by hospital medicine team attendings

CONTACTS AND LOCATIONS:
Overall Officials: Alvin R Rajkomar, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Patel S, Rajkomar A, Harrison JD, Prasad PA, Valencia V, Ranji SR, Mourad M. Next-generation audit and feedback for inpatient quality improvement using electronic health record data: a cluster randomised controlled trial. BMJ Qual Saf. 2018 Sep;27(9):691-699. doi: 10.1136/bmjqs-2017-007393. Epub 2018 Mar 5. PMID 29507124